CLINICAL TRIAL: NCT07013695
Title: Evaluation of the Impact of Virtual Reality on Sedation Use in Patients Undergoing Regional Anesthesia for Scheduled Orthopedic Surgery
Acronym: VIRTUALR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Eure-Seine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A00055-38
Record Dates: First submitted 2025-05-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Orthopedic Procedure; Anesthesia; Sedation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized parallel-group study with two arms (virtual reality group vs. control group) comparing the effect of virtual reality on sedation use during regional anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality group (Active Comparator): Participants in this group receive a virtual reality session with a hypnotic objective during surgery performed under regional anesthesia. The device consists of a virtual reality headset offering immersive visual and auditory content in a calming environment chosen by the participant. The session begins before the administration of regional anesthesia and may continue throughout the surgical procedure.
  Interventions: Device: Virtual reality headset
- Control Group (Placebo Comparator): Participants in this group receive standard anesthetic and surgical care without the use of virtual reality.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Device: Virtual reality headset — Patients in the intervention group receive a virtual reality session with a hypnotic purpose during surgery under regional anesthesia. The device consists of a virtual reality headset providing visual and auditory immersion in a calming environment, freely chosen by the patient. The session begins before the regional anesthesia is administered and may continue throughout the entire surgical procedure
  Arms: virtual reality group
Other: Standard Care (in control arm) — Participants in this group receive standard anesthetic and surgical care without the use of virtual reality
  Arms: Control Group

SUMMARY:
The VIRTUALR study evaluates the effect of virtual reality combined with hypnosis on anxiety in patients undergoing orthopedic surgery under regional anesthesia. Patients are randomly assigned to two groups: one group receiving virtual reality and a control group without the device. Anxiety and satisfaction questionnaires are used to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient affiliated with or benefiting from a social security system
* Patient aged 18 years or older
* Patient requiring regional anesthesia for scheduled orthopedic surgery of the upper or lower limb

Exclusion Criteria:

* Patient refusal to participate in the study
* Device interfering with the surgical or anesthetic procedure
* Premedication before arrival in the operating room
* Psychiatric or cognitive disorders, communication disorders
* Patient unable to understand the study (language barrier, psychological issues)
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-07-17 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
Comparison of sedation use rates between the experimental group and the control group (level 0 versus ≥1). | Intraoperative period (from arrival in the operating room to the end of surgery)
  Proportion of patients who required sedation (at level ≥1) during regional anesthesia or surgery, compared to those who did not receive sedation (level 0). Sedation levels are defined according to a standardized scale.

SECONDARY OUTCOMES:
Mean age of patients | Baseline (before anesthesia consultation or at inclusion)
  Mean age of patient in each group at baseline
Sex distribution | Baseline (before anesthesia consultation or at inclusion)
  Number of male and female patients in each group
type of surgery | Baseline (before anesthesia consultation or at inclusion)
  Distribution of types of surgery performed in each group
ASA score distribution | Baseline (before anesthesia consultation or at inclusion)
  Distribution of ASA physical status scores among patients in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste HARDY, Principal Investigator — Centre Hospitalier Eure-Seine
Locations (1):
- Centre Hospitalier Eure-Seine, Évreux, France

IPD SHARING:
Plan to Share IPD: No